CLINICAL TRIAL: NCT00652210
Title: Use of Multiphoton Microscopy in the Diagnosis of Cancer
Acronym: MPM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Douglas S. Scherr, Associate Professor, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0506007919
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Bladder Cancer; Prostate Cancer
Keywords: Bladder cancer; prostate cancer; multiphoton microscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms | interventions — Microscopy, Fluorescence, Multiphoton

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MPM (Experimental): Subject tissue was reviewed using multiphoton microscopy
  Interventions: Other: Multiphoton microscopy

INTERVENTIONS:
Other: Multiphoton microscopy — Use of multiphoton microscopy to diagnose cancer

SUMMARY:
Multiphoton microscopy (MPM) has been shown to be able to image tissue at a cellular level. Our project will initially evaluated the ability of MPM imaging to distinguish normal bladder urothelium from atypical and malignant urothelium in the ex vivo setting. After development of sufficient criteria, we plan to develop an endoscopic bladder probe that will provide a non-invasive means to image the interior of the bladder at the cellular level, which would provide direct evidence of the presence of tumor without a biopsy. After exhibiting usefulness of MPM imaging for bladder cancer, we will look at other organs beginning with the colon.

DETAILED DESCRIPTION:
Same as above

ELIGIBILITY:
Inclusion Criteria:

* Anyone who presents with bladder and/or prostate cancer

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2005-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
After several delays, the multiphoton microscope has been delivered to Weill Cornell Medical College. We have been using this time to set-up and fine tune the multiphoton microscope. As of current, no negative events have occurred. | 10/14/2007 to 2/15/2008

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Scherr, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States